CLINICAL TRIAL: NCT02037399
Title: Pilot Trial on Efficacy of Single Dose Perioperative Intravenous Dexamethasone for Pain Relief After Endoscopic Submucosal Dissection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0577
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Early Gastric Cancer or Gastric Adenoma
Keywords: Endoscopic submucosal dissection; early gastric cancer; pain relief; intravenous dexamethasone; present pain intensity
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intravenous dexamethasone (Experimental): To receive intravenous dexamethasone (0.15 mg/kg) immediately after ESD
  Interventions: Drug: intravenous dexamethasone
- intravenous normal saline (Placebo Comparator): To receive normal saline as placebo intravenous immediately after ESD
  Interventions: Drug: intravenous normal saline

INTERVENTIONS:
Drug: intravenous dexamethasone — Patients were enrolled in outpatient settings after evaluating appropriate ESD indications. A single study coordinator performed a randomization process by using a table of random numbers. The patients were allocated to receive intravenous dexamethasone (0.15 mg/kg) immediately after ESD. The patients with an odd number were assigned into DEXA group, and the patients with an even number were assigned into placebo group. The syringe including dexamethasone was completely covered with a paper sticker to mask treatment assignment. The operator and assisting nurse were also blinded to the study.
  At the day and next day of ESD, intravenous proton pump inhibitor was routinely administered to prevent complications including bleeding. At 3rd day of ESD, all patients started to take 40mg oral lansoprazole once a day and sucralfate suspension 3 times a day for 28 days.
  Arms: intravenous dexamethasone
Drug: intravenous normal saline — Patients were enrolled in outpatient settings after evaluating appropriate ESD indications. A single study coordinator performed a randomization process by using a table of random numbers. The patients were allocated to receive intravenous normal saline as placebo immediately after ESD. The patients with an odd number were assigned into DEXA group, and the patients with an even number were assigned into placebo group. The syringe including placebo was completely covered with a paper sticker to mask treatment assignment. The operator and assisting nurse were also blinded to the study.
  At the day and next day of ESD, intravenous proton pump inhibitor was routinely administered to prevent complications including bleeding. At 3rd day of ESD, all patients started to take 40mg oral lansoprazole once a day and sucralfate suspension 3 times a day for 28 days.
  Arms: intravenous normal saline

SUMMARY:
Besides major ESD-related complications, minor adverse events after ESD are also commonly noticed. Pain is one of minor ESD-related complications. . The causes of pain associated with ESD or gastric polypectomy are thought to be associated with transmural burn or transmural air leak. How control localized pain for patients who suffered from pain after ESD is appearing as new medical interests. There are few studies about management strategy for pain after ESD. Glucocorticoids are used to reduce inflammation and tissue damage in various clinical settings including inflammatory disease, rheumatic disease, and so on. The efficacy of glucocorticoids for reducing pain after surgery has recently been investigated. Glucocorticoids are thought to locally inhibit collagen deposition and fibrosis and finally reduce scar-tissue formation. Especially systemic steroids are easy to achieve a continuous effect through stable serum concentrations. If pain was partially associated with acute inflammation, we assumed intravenous dexamethasone could be helpful to relieve pain after ESD based on previous studies. we aimed to assess the efficacy of single dose postoperative intravenous dexamethasone for pain relief after ESD.

ELIGIBILITY:
Inclusion Criteria:

* 20 years of age or older
* pathologically diagnosed gastric adenoma or cancer that was eligible for ESD
* patients who gave written informed consent from patients or responsible family members.

Exclusion Criteria:

* patients who take pain killer within 48 hours or regularly at enrollment
* confirmed any other disease which can induce epigastric pain such as peptic ulcer disease and gastroesophageal reflux disease
* multiple gastric lesions for ESD
* history of gastric surgery at enrollment
* severe underlying disease including infection, cardiopulmonary disease, and diabetes.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
present pain intensity (PPI) | at 6 hours after ESD
  The primary outcomes of this study was present pain intensity (PPI) measured at 6 hours after ESD. The reason for adopting 6- hour PPI as primary endpoint was due to maximized pain at 6 hours after ESD in our pilot study.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Worni M, Schudel HH, Seifert E, Inglin R, Hagemann M, Vorburger SA, Candinas D. Randomized controlled trial on single dose steroid before thyroidectomy for benign disease to improve postoperative nausea, pain, and vocal function. Ann Surg. 2008 Dec;248(6):1060-6. doi: 10.1097/SLA.0b013e31818c709a. PMID 19092351
- [Background] Diakos EA, Gallos ID, El-Shunnar S, Clarke M, Kazi R, Mehanna H. Dexamethasone reduces pain, vomiting and overall complications following tonsillectomy in adults: a systematic review and meta-analysis of randomised controlled trials. Clin Otolaryngol. 2011 Dec;36(6):531-42. doi: 10.1111/j.1749-4486.2011.02373.x. PMID 21812940
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397
- [Background] Kiriyama S, Oda I, Nishimoto F, Mashimo Y, Ikehara H, Gotoda T. Pilot study to assess the safety of local lidocaine injections during endoscopic submucosal dissection for early gastric cancer. Gastric Cancer. 2009;12(3):142-7. doi: 10.1007/s10120-009-0514-y. Epub 2009 Nov 5. PMID 19890693